CLINICAL TRIAL: NCT02541019
Title: Prophylactic Antiemetic Efficacy of Palonosetron Versus Ondansetron for the Prophylaxis of Postoperative Nausea and Vomiting (PONV) in Women Over 60 Years Undergoing Laparoscopic Cholecystectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Federal de Bonsucesso (Other)
Responsible Party: Principal Investigator, Estevão Braga, Md, Hospital Federal de Bonsucesso
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 48149215.0.0000.5253
Record Dates: First submitted 2015-08-25; First posted 2015-09-04 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: C23.888.821.712.700
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Ondansetron; Palonosetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Palonosetron (Experimental): Palonosetron (iv) one minute before anesthesic induction.
  Interventions: Drug: Palonosetron
- Ondansetron (Experimental): ondansetron (iv) one minute before anesthesic induction and ondansetron regular three times a day for two days after the surgery.
  Interventions: Drug: Ondansetron

INTERVENTIONS:
Drug: Ondansetron — 4 mg IV, one minute before the anesthesia induction and 4 mg IV three times a day during two days after the surgery.
  Arms: Ondansetron
Drug: Palonosetron — 75 mcg IV, one minute before the anesthesia induction.
  Arms: Palonosetron

SUMMARY:
Despite the development of new drugs, nausea and vomiting after surgery (PONV) are still frequent. Antagonists 5HT3 receptors, such as ondansetron and palanosetron, are among the main characterized prophylactic agents in patients at high risk, however there are few studies comparing the efficacy of these drugs and no study that addresses women aged over 60 years.

In this prospective, randomized, double-blind study, 80 women nonsmokers, undergoing laparoscopic cholecystectomy will be divided into two groups, receiving during anesthetic induction intravenous ondansetron 4 mg (n = 40) or palonosetron 75 mcg (n = 40) prophylaxis of PONV.

DETAILED DESCRIPTION:
Clinical, prospective, randomized double-blind trial will be conducted at the Federal Hospital Bonsucesso (HFB), Rio de Janeiro, Brazil. Eighty female patients, olther than 60 years, ASA I to III, undergoing laparoscopic cholecystectomy will be studied. They will be randomized into two groups of 40. One group will receive Palonosetron 75 mcg (Group P) and the other will receive Ondansetron 4mg (Group O). Patients will not receive premedication. Will be monitored in the operating room with non-invasive blood pressure, cardioscopy, pulse oximetry, capnography and bispectral index (BIS). After cannulation of peripheral vein, 10 ml of blood will be collected for further analysis. They will be given one minute before induction of anesthesia, intravenous (IV) bolus preparations of the studied antiemetics. Patients will be pre-oxygenated with oxygen at 100% for 5 minutes and the anesthetic induction is performed with intravenous administration of fentanyl 3 mcg / kg; Lidocaine 1.5 mg / kg and propofol 2 mg / kg. Tracheal intubation will be facilitated after 3 minutes of administration of Rocuronium 0.6 mg / kg EV .Maintenance of anesthesia will be with Sevoflurane 2 L / min in 50% oxygen / air, with its concentration adjusted to maintain BIS between 40-60. Remifentanil 0.05 mcg / kg / min to 0.2 mcg / kg / min IV can be administered intraoperatively if the heart rate or blood pressure to rise more than 20% of values baseline. Additional doses of rocuronium may also be administered as needed. Patients will receive paracoxibe 40 mg,dipirone 50 mg / kg and 50 mg of ranitidine IV after tracheal intubation and have the surgical wound infiltration with 20 mL of ropivacaine 0.5%, before the sutures. Neuromuscular blockade reversed with neostigmine 0.04 mg / kg and atropine 0.02 mg / kg IV at the end of surgery. Will be limited to insufflation of the pneumoperitoneum to abdominal pressure of 15 mmHg.

A non-participating physician will be aware of the research on which antiemetic was given and be responsible for postoperative prescription of patients. The researchers did not have access to prescription and medical records within 48 hours after surgery. Both groups will recive metoclopramide 10 mg (EV) as rescue medication for PONV, and the Group O will continue with prescription ondansetron 4 mg (EV) regular 8 / 8h, in the following 48 h after surgery. Patients will receive clinical visit by the research team 2, 6, 24 and 48 h after the end of surgery and will be questioned about the frequency and intensity of PONV, as well as other side effects. Finished the last evaluation, researchers will review the prescription and will note the use of opioids (type, dose, route of administration), use of rescue medication, total cost of antiemetic therapy (including 5HT3 antagonist and rescue medication), based on "Brasíndice" table.

All patients have their blood samples analyzed in the clinical research laboratory of the Universidade Federal Fluminense, for concurrent research of prevalence of polymorphisms of 5HT3 receptors and their correlation with the antiemetic effect. DNA will be extracted from blood samples using a kit to genomic DNA purification. Polymerase chain reaction test for real time will be applied below for analysis of single nucleotide polymorphisms of. The reactions are prepared with Genotyping according to the manufacturer's instructions and performed on a sequence detection system using standard thermal cycling conditions.

ELIGIBILITY:
Inclusion Criteria:

* Will be selected patients aged over 60 years, ASA 1-3 that are candidates for laparoscopic cholecystectomy

Exclusion Criteria:

* Participation in another study last month.
* Body mass index> 35.
* The occurrence of episodes of nausea or vomiting in the last 24 h prior to surgery.
* Use of corticosteroids.
* Smoking.
* Alcoholism.
* Use of psychoactive drugs or any other drug with antiemetic effect.
* Known hypersensitivity to any study medication
* Severe diseases in organs such as kidney, liver, lung, heart, brain and bone marrow.
* Conversion laparoscopic cholecystectomy for conventional cholecystectomy.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-10; Primary Completion 2017-01-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Frequency and intensity of individual episodes of PONV. | 48 h after surgery

SECONDARY OUTCOMES:
Intensity of nausea | during clinical visit 2, 6, 24 and 48 h postoperatively
  Evaluate nausea intensity in numeric scale (0-10) during clinical visit
Need of medication for antiemetic rescue | during the 48 h after surgery
  Assess the need of medication for antiemetic rescue during the 48 h after surgery
Number of complete responders to medication | during the 48 h after surgery
  Determine the number of complete responders to medications (no emetic episode or rescue medication during the 48 hours after surgery)
Degree of satisfaction with antiemetic therapy | during the 48 h after surgery
  Know the degree of satisfaction with antiemetic therapy, through the 5-point rating scale (very dissatisfied, dissatisfied, neutral, satisfied or very satisfied)
Cost of antiemetic medication | during the 48 h after surgery
  total cost of antiemetic therapy (including 5HT3 antagonist and rescue medication), based on the table "Brasíndice".
Frequency and intensity of adverse effects | during the 48 h after surgery
  Determine the frequency and intensity of adverse effects by means of numerical scale(0-10) (headache, dizziness, drowsiness and others)
Frequency of polymorphism of 5HT3a receptors and 5HT3b | participants will be followed for the duration of hospital stay, an expected average of 48 h
  To assess the frequency of polymorphism and 5HT3b 5HT3a receptors and their correlation with the frequency and intensity of antiemetic effect and adverse effects.

CONTACTS AND LOCATIONS:
Overall Officials: Ismar L Cavalcanti, PhD, Principal Investigator — UFF
Locations (1):
- Hospital Federal de Bonsucesso, Rio de Janeiro, Brazil

REFERENCES:
- [Result] Horn CC, Wallisch WJ, Homanics GE, Williams JP. Pathophysiological and neurochemical mechanisms of postoperative nausea and vomiting. Eur J Pharmacol. 2014 Jan 5;722:55-66. doi: 10.1016/j.ejphar.2013.10.037. Epub 2013 Oct 26. PMID 24495419
- [Result] Silva AC, O'Ryan F, Poor DB. Postoperative nausea and vomiting (PONV) after orthognathic surgery: a retrospective study and literature review. J Oral Maxillofac Surg. 2006 Sep;64(9):1385-97. doi: 10.1016/j.joms.2006.05.024. PMID 16916674
- [Result] Grover VK, Mathew PJ, Hegde H. Efficacy of orally disintegrating ondansetron in preventing postoperative nausea and vomiting after laparoscopic cholecystectomy: a randomised, double-blind placebo controlled study. Anaesthesia. 2009 Jun;64(6):595-600. doi: 10.1111/j.1365-2044.2008.05860.x. PMID 19453311
- [Result] Turkistani A, Abdullah K, Manaa E, Delvi B, Khairy G, Abdulghani B, Khalil N, Damas F, El-Dawlatly A. Effect of fluid preloading on postoperative nausea and vomiting following laparoscopic cholecystectomy. Saudi J Anaesth. 2009 Jul;3(2):48-52. doi: 10.4103/1658-354X.57872. PMID 20532102
- [Result] Oksuz H, Zencirci B, Ezberci M. Comparison of the effectiveness of metoclopramide, ondansetron, and granisetron on the prevention of nausea and vomiting after laparoscopic cholecystectomy. J Laparoendosc Adv Surg Tech A. 2007 Dec;17(6):803-8. doi: 10.1089/lap.2006.0243. PMID 18158814
- [Result] Rusch D, Eberhart LH, Wallenborn J, Kranke P. Nausea and vomiting after surgery under general anesthesia: an evidence-based review concerning risk assessment, prevention, and treatment. Dtsch Arztebl Int. 2010 Oct;107(42):733-41. doi: 10.3238/arztebl.2010.0733. Epub 2010 Oct 22. PMID 21079721
- [Result] Rueffert H, Thieme V, Wallenborn J, Lemnitz N, Bergmann A, Rudlof K, Wehner M, Olthoff D, Kaisers UX. Do variations in the 5-HT3A and 5-HT3B serotonin receptor genes (HTR3A and HTR3B) influence the occurrence of postoperative vomiting? Anesth Analg. 2009 Nov;109(5):1442-7. doi: 10.1213/ane.0b013e3181b2359b. Epub 2009 Aug 27. PMID 19713259
- [Result] Janicki PK, Sugino S. Genetic factors associated with pharmacotherapy and background sensitivity to postoperative and chemotherapy-induced nausea and vomiting. Exp Brain Res. 2014 Aug;232(8):2613-25. doi: 10.1007/s00221-014-3968-z. Epub 2014 May 4. PMID 24792505
- [Result] Trammel M, Roederer M, Patel J, McLeod H. Does pharmacogenomics account for variability in control of acute chemotherapy-induced nausea and vomiting with 5-hydroxytryptamine type 3 receptor antagonists? Curr Oncol Rep. 2013 Jun;15(3):276-85. doi: 10.1007/s11912-013-0312-x. PMID 23512709
- [Result] Choi YS, Shim JK, Yoon DH, Jeon DH, Lee JY, Kwak YL. Effect of ramosetron on patient-controlled analgesia related nausea and vomiting after spine surgery in highly susceptible patients: comparison with ondansetron. Spine (Phila Pa 1976). 2008 Aug 1;33(17):E602-6. doi: 10.1097/BRS.0b013e31817c6bde. PMID 18670328
- [Result] Apfel CC, Roewer N. Risk assessment of postoperative nausea and vomiting. Int Anesthesiol Clin. 2003 Fall;41(4):13-32. doi: 10.1097/00004311-200341040-00004. No abstract available. PMID 14574212